CLINICAL TRIAL: NCT04409171
Title: Alteration of Glucose Metabolism After Partial Pancreatectomy Assessed With Biochemical Markers :A Single Center Prospective Observational Study
Brief Title: Glucose Metabolism After Partial Pancreatectomy
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yoo-Seok Yoon, Associate Professor, Seoul National University Bundang Hospital
Other Study IDs: SNUBH-GS-HBP6
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Pancreatectomy; Hyperglycemia; Diabete Mellitus
Keywords: Pancreatectomy; Diabetes Mellitus; pancreaticoduodenectomy
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD: pancreaticoduodenectomy
  Interventions: Diagnostic Test: oral glucose tolerance test
- DP: distal pancreatectomy
  Interventions: Diagnostic Test: oral glucose tolerance test

INTERVENTIONS:
Diagnostic Test: oral glucose tolerance test

SUMMARY:
This is a single center observational study to assess alteration of glucose metabolism after pancreatectomy.

DETAILED DESCRIPTION:
Biochemical markers of glucose metabolism including oral glucose tolerance tests, fasting blood glucose, insulin, glucagon and HbA1c were performed on patients receiving pancreatectomy (pancreaticoduodenectomy and distal pancreatectomy). Tests were done preoperatively, postoperatively at 3 months, and at 1 year. The primary endpoints were the incidence and risk factors of new-onset and worsened DM after each type of pancreatectomy.

ELIGIBILITY:
Inclusion Criteria:

* partial pancreatectomy

Exclusion Criteria:

* total pancreatectomy
* incomplete testing
* follow-up loss
* death within 1 year

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients receiving partial pancreatectomy
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
incidence & risk factors of new-onset DM | at 1 year
  incidence & risk factors of new onset DM after pancreatectomy
incidence & risk factors of worsened DM | at 1 year
  incidence & risk factors of worsened DM after pancreatectomy

SECONDARY OUTCOMES:
characteristics of new-onset and worsened DM | 1 year
  changes of glucose metabolism during study period

IPD SHARING:
Plan to Share IPD: No
There are no plans of sharing IPD

REFERENCES:
- [Background] Lee BW, Kang HW, Heo JS, Choi SH, Kim SY, Min YK, Chung JH, Lee MK, Lee MS, Kim KW. Insulin secretory defect plays a major role in the development of diabetes in patients with distal pancreatectomy. Metabolism. 2006 Jan;55(1):135-41. doi: 10.1016/j.metabol.2005.08.005. PMID 16324932
- [Background] Hwang HK, Park J, Choi SH, Kang CM, Lee WJ. Predicting new-onset diabetes after minimally invasive subtotal distal pancreatectomy in benign and borderline malignant lesions of the pancreas. Medicine (Baltimore). 2017 Dec;96(51):e9404. doi: 10.1097/MD.0000000000009404. PMID 29390555